CLINICAL TRIAL: NCT07098468
Title: Evaluation of the Incidence and Risk Factors of Myocardial Injury After Noncardiac Surgery (MINS) in Patients Undergoing Knee and Hip Arthroplasty
Brief Title: Myocardial Injury After Noncardiac Surgery (MINS) in Patients Undergoing Knee and Hip Arthroplasty
Acronym: MINS
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Mehmet sahap, Asist prof, Ankara City Hospital Bilkent
Other Study IDs: MINS
Record Dates: First submitted 2025-07-14; First posted 2025-08-01 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: MYOCARD INFARCTUS; Non Cardiac Surgery; ARTHROPLASTY, REPLACEMENT; ANESTHESIA
Keywords: Myocardial injury, noncardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 180 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mins positivity: Patients with high sensitive troponin positivity after surgery
- Mins Negative: Patients with negative high sensitive troponin after surgery

SUMMARY:
The aim of this study is to determine the incidence of myocardial injury after noncardiac surgery (MINS) in patients undergoing elective total knee or hip arthroplasty, and to identify the demographic, clinical, laboratory, and surgical risk factors that may contribute to its development.

DETAILED DESCRIPTION:
Cardiovascular complications that develop during the perioperative period stand out as a significant cause of morbidity and mortality in patients after surgery. Especially myocardial injury (MINS) occurring after non-cardiac surgeries often progresses without clinical symptoms and signs, and therefore its diagnosis can be missed. The early detection of this silent damage is of great importance for patient safety and treatment management. It is reported that 5% to 25% of patients after non-cardiac surgery have elevated cardiac troponin (cTn) levels, and most of these patients are asymptomatic. This situation suggests that many patients are exposed to undetected myocardial damage. In patients who have experienced myocardial infarction (MI) or myocardial injury, morbidity and mortality rates are high not only before surgery but also on the 30th day and even up to the 1st year. MINS is typically detected during the perioperative period through measurements of cardiac troponin I (cTnI) or cardiac troponin T (cTnT).

These proteins are the fundamental regulatory proteins of the myocardium and are sensitive and specific biomarkers for myocardial damage. Elevations in troponin levels should be identified within the first 30 days, but these elevations typically occur within the first 2 days of the postoperative period. When high-sensitivity troponin T (hs-cTnT) measurements are used, an increase of 5 ng/L or more over the previous value has been independently associated with 30-day mortality in a major international study. The aim of this study is to determine the incidence of myocardial injury after non-cardiac surgery (MINS) in patients undergoing elective total knee or hip arthroplasty and to identify the demographic, clinical, laboratory, and surgical risk factors that may contribute to it.

ELIGIBILITY:
Inclusion Criteria:

* Age over 45
* Elective total knee or hip replacement

Exclusion Criteria:

* Those undergoing cardiac surgery
* History of acute MI (<30 days)
* Chronic elevation of troponin

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is planned to include 314 patients aged 45 and older undergoing elective hip or knee arthroplasty. Participants will be accepted for participation with physician approval and a voluntary consent form.
Sampling Method: Probability Sample
Enrollment: 314 (Estimated)
Dates: Start 2025-08-03 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Ischemia-related myocardial damage after noncardiac surgery | After surgery 30 days
  Diagnostic Biochemical Criteria for MINS:
  Myocardial Injury after Non-Cardiac Surgery (MINS) is defined when at least one of the following high-sensitivity cardiac troponin T (hs-cTnT) criteria is met:
  A postoperative hs-cTnT level of at least 20 ng/L combined with a minimum absolute increase of 5 ng/L from the preoperative value, or
  An absolute postoperative hs-cTnT concentration of ≥ 65 ng/L, regardless of baseline values.
  These threshold values are used to detect subclinical myocardial injury due to ischemia that occurs after surgery, even in the absence of ischemic symptoms or electrocardiographic changes.
  In this study, patients meeting at least one of the above criteria within 30 days postoperatively will be classified as having MINS.

SECONDARY OUTCOMES:
Causes of myocardial damage due to ischemia following noncardiac surgery | 30 days
  In this study, a secondary outcome is to investigate the causes of myocardial injury due to ischemia following non-cardiac surgery. Factors such as perioperative hemodynamic instability, type and duration of surgery, pre-existing cardiovascular comorbidities, and intraoperative events will be evaluated to identify potential contributors to ischemic myocardial damage

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Şahap, Study Director — Sahap
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to the inadequate database network, patient information will not be shared with third parties. Patient data may be shared with journals upon request.